CLINICAL TRIAL: NCT01027299
Title: A Randomised Study of Temporary Epicardial Cardiac Resynchronisation Versus Conventional Right Ventricular Pacing in Cardiac Surgical Patients.
Brief Title: Temporary Epicardial Cardiac Resynchronisation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09/CAD/4628
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2011-06

CONDITIONS: Cardiac Failure
Keywords: cardiac failure; thoracic surgery; cardiac pacing, artificial
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard pacing (Active Comparator): Standard pacing settings prescribed by the cardiac surgeon or intensivist after revascularisation.
  Interventions: Device: Biventricular pacing
- BiVentricular pacing (BiV). (Active Comparator): The group of patients receiving biventricular pacing after cardiac surgery.
  Interventions: Device: Biventricular pacing

INTERVENTIONS:
Device: Biventricular pacing — Optimised temporary biventricular pacing.
  Other Names: Standard pacing

SUMMARY:
This trial will investigate the clinical and haemodynamic effects of temporary biventricular pacing after cardiac surgery. Subjects with poor left ventricular systolic function will receive either temporary biventricular pacing or 'standard' post-operative pacing for 48 hours.

The investigators hypothesis that reversal of cardiac dyssynchrony will improve tissue perfusion and cardiac haemodynamics after surgical revascularisation. This will shorten post-operative recovery in cardiac ITU.

DETAILED DESCRIPTION:
Patients with poor left ventricular (LV) function are at higher risk of complications after cardiac surgery, compared to patients with preserved LV function. The higher complication rates also lead to prolonged Cardiac Intensive Care (CITU) admissions for monitoring and multi-organ support.

The investigators hypothesise that BiV pacing will reverse cardiac dyssynchrony and improve target organ perfusion. This will be significantly reduced the post operative requirement for Level 3 CITU care.

This study will compare 48 hours of temporary biventricular (BiV) pacing to enhance cardiac function against standard post-operative pacing, in patients with poor LV function undergoing cardiac surgery. Temporary biventricular (BiV) pacing will be achieved with the addition of a third pacing electrode attached to the left ventricle. Using a pulmonary arterial catheter the interventricular (VV) delay will be adjusted to yield the maximum cardiac output at constant heart rate- sequential BiV pacing. A pilot study conducted at the University Hospital of Wales (UHW) showed that this approach is likely to be successful.

The primary endpoint of the study will be the mean duration of Level 3 CITU care required by patients after cardiac surgery. Secondary endpoints will include: haemodynamic improvement with BiV pacing; post-operative renal function; atrial fibrillation (AF)/ ventricular arrhythmias; post operative inotropic requirements and changes in biomarkers- NT Pro BNP and Troponin T.

ELIGIBILITY:
Inclusion Criteria:

* Coronary disease scheduled for surgical revascularisation. Ejection fraction <35% (simpson's method.)

Exclusion Criteria:

* Permanent pacemaker or implantable defibrillator. Dialysis dependent renal failure. Permanent atrial fibrillation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Duration of Level 3 care after cardiac surgery, as defined by the 'Designed for Life' document- Welsh Assembly Government. | 30 days

SECONDARY OUTCOMES:
Mortality | 30 days
Haemodynamic support after surgery (inotropes/ intra-aortic balloon pump.) | 30 days
Vascular event (stroke or myocardial infarction.) | 30 days
post operative arrhythmia. | 48 hours
Haemodynamic measurements of cardiac status (Pulmonary arterial catheter, echo data and FloTrac monitor). | 48 hours
Renal function and requirement for haemofiltration. | 30 days
Biomarkers (Troponin T and NT Pro BNP.) | 72 hours
Re-intubation or re-sternotomy. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Zaheer R Yousef, MD, Study Director — Cardiff and Vale Local Heath Board, Cardiff.
Locations (2):
- United Kingdom (2):
  - Cardiff and Vale University Health Board., Cardiff
  - Morriston Hospital, Swansea

REFERENCES:
- [Derived] Russell SJ, Tan C, O'Keefe P, Ashraf S, Zaidi A, Fraser AG, Yousef ZR. Optimized temporary bi-ventricular pacing improves haemodynamic function after on-pump cardiac surgery in patients with severe left ventricular systolic dysfunction: a two-centre randomized control trial. Eur J Cardiothorac Surg. 2012 Dec;42(6):e146-51. doi: 10.1093/ejcts/ezs492. PMID 23138590
- [Derived] Russell SJ, Tan C, O'Keefe P, Ashraf S, Zaidi A, Fraser AG, Yousef ZR. Temporary epicardial cardiac resynchronisation versus conventional right ventricular pacing after cardiac surgery: study protocol for a randomised control trial. Trials. 2012 Feb 20;13:20. doi: 10.1186/1745-6215-13-20. PMID 22348447